CLINICAL TRIAL: NCT05692778
Title: Optimized Care of People With Diabetes and Foot Complication in Primary Care
Status: Recruiting | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Ulla Hellstrand Tang, Principal Investigator, Sahlgrenska University Hospital
Other Study IDs: Dnr 2020-02175
Record Dates: First submitted 2023-01-07; First posted 2023-01-20 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Diabetes; Diabetic Foot; Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Diabetes Complications
Keywords: diabetes; diabetic foot; eHealth; foot deformities; prevention; co-design
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Diabetes Complications; Foot Deformities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Patients being foot examined by using an eHealth tool: Patients being foot examined by using an eHealth tool
  Interventions: Other: Patients being foot examined by using an eHealth tool
- 2: Patients being foot examined in traditional manner: Patients being foot examined in traditional manner
  Interventions: Other: Patients being foot examined in traditional manner

INTERVENTIONS:
Other: Patients being foot examined by using an eHealth tool — Patients being foot examined by using an eHealth tool that has been developed, will be tested with the intention to implement the eHealth tool
  Groups: 1: Patients being foot examined by using an eHealth tool
Other: Patients being foot examined in traditional manner — Patient are being foot examined in the way as health care professionals usually make the foot examination in patients with diabetes
  Groups: 2: Patients being foot examined in traditional manner

SUMMARY:
The goal of this observational study is to create and evaluate and new management, by using eHealth tools, to prevent diabetic foot ulcers. The main questions it aims to answer are:

1. Validation

   a. Is a method for foot assessment, that uses eHealth tools, valid regarding its usefulness? b. Is a method for foot assessment, that uses eHealth tools, reliable regarding the generated risk stratification?
2. Mapping

   1. How do health care professionals and patients with diabetes experience that the future foot examination should be designed?
   2. What experiences have health care professionals and patients with diabetes to use an eHealth tool supporting the annual foot examination?
3. Interviews - to use a paper format supporting a structured foot assessment

   a. How do health care professionals experience to use a structured foot form, in paper form?
4. Interviews - footwear

   a. What factors that influence how patients with diabetes choose their footwear?
5. Interviews - usability test of using an eHealth tool

   a. How could a digital eHealth tool be designed? b. How could a digital eHealth solution be implemented, managed and spread in public health care setting? i. Participants will:

1. fill in questionnaires 2. be interviewed 3. test eHealth solutions supporting the foot examination

6. Experiences of using an eHealth tool supporting the foot assessment

a. How could a digital eHealth tool be designed?

7. Questionnaires regarding self-perceived quality of life, the experiences of the visit at the care unit, transportation to the care unit.

a. Patients that visits care fills in a questionnaire regarding self-perceived quality of life (EQ-5D), a modified version of National Patient Survey, the diabetes questionnaire and a questionnaire regarding their travels and time for travels to and from the visit to the care unit.

8. Critical evaluation of complexity

1. Exists complexity in the development, test, management, spread and sustain of an eHealth tool supporting foot examination and self-care of the feet in diabetes.
2. How could a digital eHealth solution be implemented, managed and spread in public health care setting?

   9. Long term effect

a. What is the long-term effect of using an eHealth tools supporting a structured foot examination?

DETAILED DESCRIPTION:
1. Method - Validation

   Below is a description of the method used to answer the research questions:

   a. Is a method for foot assessment, that uses eHealth tools, valid regarding its usefulness? b. Is a method for foot assessment, that uses eHealth tools, reliable regarding the generated risk stratification? An interdisciplinary expert group will validate, in a series of meetings, what items to include in a structured foot assessment, called "D-Foot CARE" aimed to assess the risk to develop diabetic foot ulcers. Procedures, how to make the specific foot assessments in "D-Foot CARE" will be developed. The content in "D-Foot CARE" will be based on scientific literature, clinical guidelines and recommendation. The validation process is documented by the principal investigator.
2. Method - Mapping

Below is a description of the method used to answer the research questions:

1. How do health care professionals and patients with diabetes experience that the future foot examination should be designed?
2. What experiences have health care professionals and patients with diabetes to use an eHealth tool supporting the annual foot examination?

   Patients with diabetes and healthcare professionals' answers questionnaires, digital or in paper format, according to the method called Concept Mapping, a method used in action research. By using Concept mapping a variety of points of views are gathered when respondents answers an open question. Following the instructions in the survey the respondents complete a sentence. An example: "The national board of health and welfare recommends that persons with diabetes should have their feet foot checked annually. The aim is to promote good foot health. Persons with diabetes, at risk, should be treated with podiatry and be referred to the department of prosthetics & orthotics. Here, below, is an open question that you complete with your own words To improve care and self-care of the feet for persons with diabetes I suggest that….

   Information about the study is available for persons with diabetes in different ways:
   1. Through advertisement; information by the patient's organization; through primary care centers in Skaraborg and by the department of prosthetics & orthotics.
   2. At meetings arranged by the patient's organization
   3. At the primary care center Information about the study for health care professionals working with patients with diabetes having foot complications is given from the research team.

   3. Method - interview how it is to use a paper format supporting a structured foot assessment By semi-structured interviews with healthcare professionals,, that have used a structured paper format as support when they made foot examination in patients with diabetes, their experiences of working with the paper format was evaluated.

   4. Interviews - footwear By telephone semi- structured interviews with persons with diabetes factors that influence their choice of footwear is investigated.

   5. Interviews - usability test of using an eHealth tool In usability tests the use of eHealth tools supporting care and self-care of the feet is evaluated.

   6. Experiences of using an eHealth tool supporting the foot assessment Patients with diabetes and healthcare professionals report their experiences of using eHealth tool by filling in survey, e.g. the System Usability Scale.

a. How could a digital eHealth tool be designed? b. How could a digital eHealth solution be implemented, managed and spread in public health care setting? 7. Questionnaires regarding self-perceived quality of live, the experiences of the visit at the care unit, transportation to the care unit.

a. Patients that visits care fills in EQ-5D, a modified version of National Patient Survey, the diabetes questionnaire and a questionnaire regarding their travels and time for travels to and from the visit to the care unit.

8. Critical evaluation of complexity By using the NASSS CAT framework: Non-adoption, Abandonment, Scale-up, Spread, and Sustainability of health technology; CAT: complexity assessment tool) complexities are explored and managed in the development, test, management, spread and sustain of the eHealth tool.

9. Long term effect

a. What is the long-term effect of using an eHealth tools supporting a structured foot examination?

The Researchers will compare long-term outcomes from the intervention group with a comparison group consisting of medical record data of patients from a couple of primary care centers for following parameters:

2. number of patients that have had an annual foot examination 3. number of patient that had had a digital annual foot examination 4. number of patients that have a diabetic foot ulcer 5. number of patients that hat an amputation in the lower extremities 6. risk grad 7. have had podiatry 8. location for foot care (at home, mobile team)

ELIGIBILITY:
Inclusion Criteria patients:

* Persons with diabetes being treated in Region Västra Götaland
* Understand spoken and written Swedish

Exclusion Criteria:

• Not understand spoken and written Swedish

Inclusion Criteria healthcare professionals:

* Professionals working with patients with diabetes having foot complications.
* Working in Region Västra Götaland
* Understand spoken and written Swedish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Patients living in Region Västra Götaland being treated in a care unit in the same region.
  Professionals Professionalsm working in Region Västra Götaland being treating patientes in a care unit in the same region.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Validation | 2020-2021
  A valid foot examination routine is developed and presented in paper format.
Mapping | 2020-2023
  A variety of points of views are gathered regarding how the future foot care process should be managed. The method used Concept Mapping, is a methodology for mapping ideas that integrates input from multiple sources with differing expertise or interest, creates maps with multivariate data analyses that depict the composite thinking of the group, and yields data that allows for comparisons across rating criteria, stakeholder groups, different points in time, etc. to aid in targeted planning, implementation strategies, and evaluation. Group concept mapping is related to the growing interest in the role that theory plays in planning and evaluation.
Interviews - to use a paper format supporting a structured foot assessment | 2020-2023
  Experiences regarding how do health care professionals experienced it to use a structured foot form, in paper form will be gathered using qualitative content analysis, as described by Graneheim and Lundman, is considered appropriate in order inductively to focus on and describe experiences and variations on an individual level and to identify differences and similarities on a manifest and latent level. The analysis will be conducted in several steps. First, all the data will be read several times to ensure immersion in the data. All interview text will be regarded as a unit of analysis. The text will then be divided into "meaning units" that corresponded to the aim of the study. Each meaning unit will be condensed and labelled with a code. Codes are described as concrete and as close to the text as possible.
  Semi-structured interviews will be held with two focus groups and individual interviews.
Interviews - footwear | 2023-2025
  Factors are summarized regarding how patients with diabetes choose their footwear will be gathered using qualitative content analysis, as described by Graneheim and Lundman, is considered appropriate in order inductively to focus on and describe experiences and variations on an individual level and to identify differences and similarities on a manifest and latent level. The analysis will be conducted in several steps. First, all the data will be read several times to ensure immersion in the data. All interview text will be regarded as a unit of analysis. The text will then be divided into "meaning units" that corresponded to the aim of the study. Each meaning unit will be condensed and labelled with a code. Codes are described as concrete and as close to the text as possible.
  Semi-structured interviews will be held with two focus groups or individual interviews.
Interviews - usability test of using an eHealth tool | 2020-2024
  The usability lab test is usually performed in three stages: preparation/planning, actual test and follow-up . After preparation the test will be performed, in three phases: the pre-test phase, the actual test and the post-test phase. The participants will follow the tasks assigned to the test and will be encouraged to think aloud while performing the test to gather more substantial and qualitative data. After the test, the users will be debriefed, preferably using both questionnaires and interviews. In the follow-up stage, the recordings are coded and collected data are analyzed. Specific problems found are analyzed in detail and results will be reported. System Usability Scale, a test used to gather test participants' expectations/experiences when the usability test will be used (0-100 scale).
Experiences of using an eHealth tool supporting the foot assessment | 2020-2024
  Users, will reported how they expected and perceived it to use an eHealth tool supporting the foot examination evaluated with System Usability Scale (SUS). SUS is a test used to gather test participants' expectations/experiences when the usability test will be used (0-100 scale

SECONDARY OUTCOMES:
Questionnaires regarding self-perceived quality of life, the experiences of the visit at the care unit, transportation to the care unit. | 2020-2025
  Summaries regarding self-perceived quality of life, the experiences of the visit at the care unit, transportation to the care unit are made.
  Self-perceived quality of life is measured with EQ-5D, a standardised, reliable and valid measurement of health status developed by the EuroQol Group in order to provide a simple, generic measurement of health for clinical and economic appraisal. The answers kan be levelled in: 1) I have no problems…, level 2) I have slight problems…, 3) I have moderate problems…,4) I have severe problems…,5) I am unable to… Experiences of the visit at the care unit will be measured with a modified version of the national Swedish patient survey.
  Transportation to the care unit will be registered in km and hour/minutes
Critical evaluation of complexity | 2020-2025
  By using the NASSS CAT framework: Non-adoption, Abandonment, Scale-up, Spread, and Sustainability of health technology; CAT: complexity assessment tool) complexities are explored and managed in the development, test, management, spread and sustain of the eHealth tool.
Long term effect | 2023-2028
  The Researchers will compare long-term outcomes from the intervention group with a comparison group consisting of medical record data of patients from a couple of primary care centers for following parameters, measured in numbers of patients that:
  2. had an annual foot examination 3. had a digital annual foot examination 4. have a diabetic foot ulcer 5. had an amputation in the lower extremities 6. risk grad (1-4) 7. recieved podiatry and 8. location for foot care (at home, mobile team)

CONTACTS AND LOCATIONS:
Locations (1):
- Departmetn of Prosthetics & Orthotics, Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Hellstrand Tang U, Scandurra I, Sundberg L, Annersten Gershater M, Zugner R. Patients' Expectations of Evidence-Based Service at the Pharmacy Regarding Information on Self-Care of the Feet for Persons with Diabetes at Risk of Developing Foot Ulcers - A Cross-Sectional Observational Study in Sweden. Patient Prefer Adherence. 2023 Dec 27;17:3557-3576. doi: 10.2147/PPA.S435632. eCollection 2023. PMID 38169667
- [Derived] Andersson S, Scandurra I, Nystrom U, Varemo M, Hellstrand Tang U. Experiences of a Novel Structured Foot Examination Form for Patients With Diabetes From the Perspective of Health Care Professionals: Qualitative Study. JMIR Nurs. 2023 Jul 18;6:e45501. doi: 10.2196/45501. PMID 37463012